CLINICAL TRIAL: NCT04739813
Title: Phase 1 Study of Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, and Revlimid in Combination With Polatuzumab (ViPOR-P) in Relapsed/Refractory B-cell Lymphoma
Brief Title: Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, and Revlimid in Combination With Polatuzumab (ViPOR-P) in Relapsed/Refractory B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210014; 21-C-0014
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Lymphoma; Non-Hodgkin Lymphoma; Diffuse Large B-Cell Lymphoma; Burkitt Lymphoma
Keywords: Monoclonal Antibody; Dose Finding
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma | interventions — obinutuzumab; Prednisone; Lenalidomide; polatuzumab vedotin; ibrutinib; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Dose Escalation (Experimental): Venetoclax (PO) 800mg at escalating doses (2 dose levels) on days 2-14, ibrutinib (PO) 560mg on days 1-14, prednisone (PO) 100mg on days 1-7, obinutuzumab 1000mg (IV) on days 1 and 2, lenalidomide (PO) 15mg on days 1-14, and polatuzumab (IV) at escalating doses (2 dose levels) on day 2 of each 21-day cycle (maximum 6 cycles) to determine MTD of polatuzumab and venetoclax
  Interventions: Biological: obinutuzumab; Drug: prednisone; Drug: Revlimid; Biological: Polatuzumab; Drug: ibrutinib; Drug: venetoclax
- Arm 2: Dose Expansion (Experimental): Venetoclax (PO) at the MTD days 2-14, ibrutinib (PO) 560mg on days 1-14, prednisone (PO) 100mg on days 1-7, obinutuzumab 1000mg (IV) on days 1 and 2, lenalidomide (PO) 15mg on days 1-14, and polatuzumab (IV) at the MTD of each 21-day cycle (maximum 6 cycles)
  Interventions: Biological: obinutuzumab; Drug: prednisone; Drug: Revlimid; Biological: Polatuzumab; Drug: ibrutinib; Drug: venetoclax

INTERVENTIONS:
Biological: obinutuzumab — administered intravenously, days 1 and 2, at a dose of 1000 mg; every 21 days for up to 6 cycles, or until disease progression or unacceptable toxicity
Drug: prednisone — administered orally, days 1-7, at a dose of 100 mg; every 21 days for up to 6 cycles, or until disease progression or unacceptable toxicity
Drug: Revlimid — administered orally, days 1 and 14, at a dose of 15 mg; every 21 days for up to 6 cycles, or until disease progression or unacceptable toxicity
Biological: Polatuzumab — administered intravenously, on day 2, at varying doses of 1.4-1.8 mg/kg (based upon assigned dose level); every 21 days for up to 6 cycles, or until disease progression or unacceptable toxicity
Drug: ibrutinib — administered orally, days 1-14, at a dose of 560 mg; every 21 days for up to 6 cycles, or until disease progression or unacceptable toxicity
Drug: venetoclax — administered orally, days 2-14, at a dose of 800 mg; every 21 days for up to 6 cycles, or until disease progression or unacceptable toxicity

SUMMARY:
Background:

Aggressive B-cell lymphomas can be cured but people with disease that resists treatment or that returns after treatment have poor outcomes with standard therapies. Indolent B-cell lymphomas are generally incurable with standard therapy and treatment is aimed at controlling symptoms and achieving a durable remissions. Researchers want to see if a combination of drugs can help patients with both aggressive and indolent B-cell lymphomas.

Objective:

To learn if it is safe and effective to give polatuzumab along with venetoclax, ibrutinib, prednisone, obinutuzumab, and lenalidomide to people with certain B-cell lymphomas.

Eligibility:

Adults ages 18 and older with relapsed and/or refractory B-cell lymphoma who have had at least one prior cancer treatment.

Design:

Participants will be screened with:

Medical history

Physical exam

Assessment of how they do their daily activities

Blood and urine tests

Heart function test

Tissue biopsy (if needed)

Body imaging scans (may get a contrast agent through an intravenous (IV) catheter)

Participants will have a bone marrow aspiration and/or biopsy. A needle will be put into the hipbone. Bone marrow will be removed.

Participants may give blood, tissue, saliva, or cheek swab samples. They may have optional biopsies.

Screening tests will be repeated during the study.

Treatment will be given for up to 6 cycles. Each cycle lasts 21 days.

Participants will take venetoclax and prednisone tablets by mouth. They will take ibrutinib and lenalidomide capsules by mouth. They will get obinutuzumab and polatuzumab by IV infusion. They will keep a medicine diary.

Participants will visit the clinic 30 days after treatment ends. They will have follow-up visits for 5 years. If needed, they can visit their local doctor instead. They may be contacted by phone, mail, etc., for the rest of their life....

DETAILED DESCRIPTION:
Background:

* Combination chemotherapy with rituximab has been the mainstay of treatment for CD20-positive B-cell lymphomas.
* Significant advances have been made in curing aggressive B-cell lymphomas with chemoimmunotherapy, but indolent lymphomas and relapsed/refractory aggressive lymphomas remain mostly incurable with chemotherapy alone.
* Targeted therapies, aimed at disrupting key survival pathways in lymphoid malignancies, are emerging and showing significant activity in non-Hodgkin lymphoma (NHL) in both the relapsed and first-line settings.
* Mechanistically based combinations of targeted agents are likely to benefit patients who cannot tolerate or who relapse after or are refractory to standard chemoimmunotherapy.
* ViPOR-P targets major survival pathways in B-cell lymphomas including BCL-2 (apoptosis); BTK (B-cell receptor signaling and NF-kB); Cereblon (NF-kB) and CD20 with additional genotoxic stress from the anti-mitotic antibody-drug conjugate targeting CD79b, polatuzumab.

Objectives:

* To determine the maximum tolerated dose (MTD) and the safety and toxicity profile of polatuzumab and venetoclax in combination with ibrutinib, prednisone, obinutuzumab and Revlimid (lenalidomide) (ViPOR-P) in relapsed/refractory B-cell lymphomas
* To determine the complete response (CR) rate of ViPOR-P in relapsed/refractory non-GCB

DLBCL

Eligibility:

* Individuals >= 18 years of age
* ECOG performance status of <= 2
* Histologically or cytologically confirmed relapsed and/or refractory B-cell lymphoma, excluding mantle cell lymphoma (MCL) and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL)
* Adequate organ function unless dysfunction secondary to lymphoma

Design:

* Open-label, single-center, non-randomized phase 1 study
* Standard 3 + 3 design will be used to determine the MTD of polatuzumab and venetoclax in combination with ibrutinib, prednisone, obinutuzumab and Revlimid (lenalidomide) (ViPOR-P) in relapsed/refractory B-cell lymphomas
* A small expansion cohort will be treated at the MTD for a further analysis of safety and preliminary activity.
* An expansion cohort of 32 patients (including 27 new patients + 5 patients already enrolled at DL3/MTD) with non-GCB DLBCL will be treated at the MTD to determine the CR rate to ViPOR-P of this aggressive lymphoma subtype.
* Maximum 6 cycles of combination targeted therapy every 21 days.
* To explore all dose levels in the phase 1 study and to assess the CR rate in non-GCB

DLBCL patients in a dose expansion at the MTD as well as to allow for the possibility of a few screen failures and inevaluable subjects, the accrual ceiling will be set at 55 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed B-cell lymphoma confirmed by the Laboratory of Pathology, NCI, as follows:

Cohorts 1 and 2:

* Aggressive B-cell lymphoma: includes DLBCL and subtypes, transformed lymphoma, Burkitt lymphoma, as well as high-grade B-cell lymphoma with MYC and/or BCL2 and/or BCL6 rearrangement(s).
* Indolent B-cell lymphoma: with the following exceptions:

  * MCL is excluded given increased risk of tumor lysis syndrome (TLS) with venetoclax compared to other non-Hodgkin lymphomas and need for venetoclax ramp-up, dose-escalation.
  * CLL/SLL is excluded given alternative dosing of FDA-approved venetoclax for relapsed CLL/SLL and increased risk of TLS with CLL/SLL compared to other non-Hodgkin lymphomas.

Cohort 3:

-Non-GCB DLBCL: includes DLBCL NOS and subtypes, transformed lymphoma, THRLBCL, as well as high-grade B-cell lymphoma with MYC and/or BCL6 rearrangement(s).

NOTE: Patients with known active CNS lymphoma are not eligible.

* Relapsed and/or refractory disease after at least 1 prior treatment regimen, as follows:

  * Aggressive B-cell lymphoma: relapsed after and/or refractory to at least 1 prior anthracycline-containing regimen
  * Indolent B-cell lymphoma: relapsed after and/or refractory to at least 1 prior anti- CD20 antibody-containing regimen.
* Patients must have evaluable disease by clinical exam (i.e., palpable lymphadenopathy, measurable skin lesions, etc.), laboratory assessment (i.e., lymphoma involvement of bone marrow or peripheral blood by morphology, cytology or flow cytometry), and/or imaging (measurable lymph nodes or masses on CT or MRI and/or evaluable FDG-avid lesions on PET).

NOTE: Lesions that have been irradiated cannot be included in the tumor assessment unless unequivocal tumor progression has been documented in these lesions after radiation therapy.

-Age >=18 years

NOTE: Because no dosing or adverse event data are currently available on the use of polatuzumab in combination with venetoclax, ibrutinib, obinutuzumab, prednisone and Revlimid(R) in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.

* ECOG performance status <=2.
* Adequate organ and marrow function as defined below unless dysfunction is secondary to lymphoma:

  * absolute neutrophil count* >=1,000/mcL
  * hemoglobin* >=8 g/dL
  * Platelets >=75,000/mcL
  * INR <=1.5 X institutional upper limit of normal (ULN) for patients not receiving therapeutic anticoagulation
  * PTT/aPTT <=1.5 X institutional ULN normal except if, in the opinion of the investigator, the aPTT is elevated because of a positive Lupus Anticoagulant, or a significant bleeding risk has been ruled out in the absence of a positive Lupus Anticoagulant
  * total bilirubin <=1.5 X institutional ULN (or <=3 X institutional ULN for patients with documented Gilberts syndrome identified by an isolated unconjugated hyperbilirubinemia in the absence of other signs of liver dysfunction and/or UGT1A1 mutational testing)
  * AST(SGOT)/ALT(SGPT) <=3 X institutional ULN
  * Serum creatinine <=2.0 mg/dL OR
  * Creatinine clearance >=30 mL/min/1.73 m2 for patients with creatinine levels above 2 mg/dL

NOTE: Cr Cl will be calculated with the use of the 24-hour creatinine clearance or eGRF in the clinical lab

* RBC transfusions and use of G-CSF will be allowed in order to meet eligibility parameters.

  * Immune-modulating drugs (IMiDs) including Revlimid(R) are known to be teratogenic and potential embryo-fetal harm can be seen with use of polatuzumab, venetoclax and ibrutinib. The effects of obinutuzumab on the developing human fetus is unknown. For these reasons, individuals of child-bearing potential and individuals able to father a child must agree to use adequate contraception as described below.

    * For individuals of childbearing potential:

      * Agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year as outlined below.
      * Agreement to refrain from donating eggs during timelines specified below.
      * Individuals of childbearing potential (ICBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to prescribing Revlimid(R) for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMSTM) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Revlimid(R) ICBP must also agree to ongoing pregnancy testing.
      * An individual is considered to be of childbearing potential if that person is post-menarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
      * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
      * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * For individuals able to father a child:

      * Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:
      * With partners of childbearing potential, individuals able to father a child must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year as noted below. Individuals must refrain from donating sperm during this same period.
      * With pregnant partners, individuals must remain abstinent or use a condom as noted below to avoid exposing the embryo.
      * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Contraception Requirements

    * Time frame/Study Drug (Pre-Treatment/During Treatment) - Individuals of childbearing potential (Time frame prior to/during dosing) / Individuals able to father a child (Time frame prior to/during dosing):

      ---All drugs; Begins 28 days prior to treatment; Begins on day 1
    * Time frame/Study Drug (Post-Treatment) - Individuals of childbearing potential (Time frame after the last dose) / Individuals able to father a child (Time frame after the last dose):

      * Venetoclax - 90 days / 90 days
      * Ibrutinib - 3 months / 3 months
      * Obinutuzumab - 18 months / 6 months
      * Revlimid(R) - 28 days / 28 days
      * Polatuzumab - 3 months / 5 months
  * All study participants must be registered into the mandatory Revlimid REMSTM program and be willing and able to comply with the requirements of Revlimid REMSTM. NOTE: Individuals of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMSTM program.
  * Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* The following restrictions apply to current or prior anti-cancer treatment, prior to the first dose of study drug:

  * Patients who are actively receiving any other investigational agents.
  * Any chemotherapy or anti-cancer antibodies within 2 weeks. NOTE: Short courses of corticosteroids or palliative XRT prior to enrollment are permitted within the 2- week washout period.
  * Radio- or toxin-immunoconjugates within 10 weeks.
  * Previous treatment with more than one of the study agents (i.e., polatuzumab, venetoclax, ibrutinib, or Revlimid(R)), excluding prior prednisone or anti-CD20 antibody treatment.
  * Prior allogeneic stem cell (or other organ) transplant within 6 months or any evidence of active graft-versus-host disease or requirement for immunosuppressants within 28 days.
  * Not recovered (i.e., <= Grade 1 or baseline) from adverse events due to previously administered anti-cancer treatment, surgery, or procedure. NOTE: Exceptions to this include events not considered to place the subject at unacceptable risk of participation in the opinion of the PI (e.g., alopecia).
* Patients requiring the use of warfarin are excluded because of potential drug-drug interactions that may potentially increase the exposure of warfarin.
* Patients requiring the following agents to the first dose of venetoclax or ibrutinib are excluded, as noted:

  * Strong CYP3A inhibitors within 7 days
  * Strong CYP3A inducers within 7 days

NOTE: Moderate CYP3A inhibitors and inducers should be used with caution and an alternative medication used, whenever possible.

* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the patient at the discretion of the investigator:

  * Symptomatic congestive heart failure, unstable angina pectoris, or uncontrolled cardiac arrhythmia
  * Uncontrolled and/or symptomatic thyroid disease
  * Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 2 weeks prior to Cycle 1, Day 1;
  * Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis; as well as active infection with HBV or HCV:

    * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
    * Patients with occult or prior HBV infection (defined as positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (HBcAb) and with negative HBsAg) may be included if HBV DNA is undetectable (i.e., none detected in copies/mL or IU/mL). These patients must be willing to undergo HBV DNA testing during treatment and in surveillance for at least 12 months after completion of study therapy.
  * Malabsorption syndrome or other condition that precludes enteral route of administration
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant individuals, or individuals who intend to become pregnant during the study, are excluded from this study because Revlimid(R) has known teratogenic effects and polatuzumab, venetoclax, ibrutinib and obinutuzumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, nursing should be discontinued if the individual is treated on study.
* HIV-positive patients are ineligible because of the potential for pharmacokinetic interactions with venetoclax, ibrutinib and Revlimid(R) and combination antiretroviral therapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Evidence of active tumor lysis syndrome based on laboratory assessment
* History of recent major surgery within 6 weeks prior to the start of Cycle 1, Day 1 other than for diagnosis
* History of other active malignancy that could affect compliance with the protocol or interpretation of results

  * Patients with a history of curatively treated basal or squamous cell carcinoma or stage 1 melanoma of the skin as well as any in situ carcinoma are eligible.
  * Patients with a malignancy that has been treated with curative intent will also be eligible. Individuals in documented remission who are not receiving active treatment prior to enrollment may be included at the discretion of the investigator.
* Known allergy to both xanthine oxidase inhibitors and rasburicase; or, known hypersensitivity to any of the study drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2031-04-04 (Estimated)

PRIMARY OUTCOMES:
Number and grade of adverse events | 21 days
  Number and grade of adverse events
Complete response (CR) rate | every 42 days for 3 assessments (e.g., every 2 cycles) and/or end of treatment
  Response rate based on Lugano Classification Response Criteria

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed every 3-6months
  time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed every 3-6months
Duration of Response (DOR) | For ORR-time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed every 3-6months, For CR-time measurement criteria are met for CR
  For ORR-time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed every 3-6months, For CR-time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed every 3-6months
Progression-free survival (PFS) | time from date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first, assessed every 3-6 months
  time from date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first, assessed every 3-6 months
Event-free survival (EFS) | time from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), or death, whichever occurs first, assessed every 3-6 months
  time from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), or death, whichever occurs first, assessed every 3-6 months
Overall survival (OS) | time from the date of study enrollment until death from any cause, assessed every 3-6 months
  time from the date of study enrollment until death from any cause, assessed every 3-6 months
Complete response (CR) rate | time measurement criteria are met for CR until the first date that progressive disease is objectively documented or death, assessed every 3-6months
  time measurement criteria are met for CR until the first date that progressive disease is objectively documented or death, assessed every 3-6months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Melani, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP. @@@@@@@@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.@@@@@@@@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0014.html